CLINICAL TRIAL: NCT02324803
Title: Phase II Study of Pazopanib as Second-line Treatment After Sunitinib in Metastatic Renal Cell Carcinoma (mRCC) Patients
Brief Title: Phase II Study of Pazopanib as Second-line Treatment After Sunitinib in mRCC Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern China Urology Cancer Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUCC001
Record Dates: First submitted 2014-12-13; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Self Efficacy; Adverse Drug Event; Carcinoma, Renal Cell
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- pazopanib once daily (Experimental): Patients received continuous treatment of 800 mg pazopanib once daily until disease progression, unacceptable toxicity, or withdrawal of consent occurred. Dose reductions by 400 mg to a lowest dose of 200 mg daily were allowed on the basis of tolerability and according to protocol-defined guidelines.
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — continuous treatment of 800 mg pazopanib once daily until disease progression
  Other Names: Votrient

SUMMARY:
assess the activity and toxicity of second-line treatment with pazopanib after failure of first-line sunitinib treatment in patients with clear cell mRCC; to investigate the potential association of DLL4, Notch1, VEGFA, PDGFRB, HIF-1α and HIF-2α with clinical response to pazopanib in mRCC patients.

DETAILED DESCRIPTION:
The primary end point was progression-free survival (PFS). Secondary end points were overall survival (OS), objective response rate (ORR) and safety. We assessed the tumor response according to the RECIST 1.1.

Efficacy was evaluated by computed tomography with contrast of the chest, abdomen, and pelvis. We performed tumor assessments with the use of imaging studies at baseline and every six weeks until the end of treatment. We also used such assessments to confirm a response (at least 4 weeks after initial documentation) and whenever disease progression was suspected. All imaging scans were evaluated by an independent imaging-review committee (IRC) blinded to study treatment. Patients who had inadequate data for study assessment was regarded as nonevaluable.

Adverse events were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Safety was assessed by physical examination and laboratory tests. Electrocardiograms (ECGs) were performed at baseline and every six weeks until the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Diagnosis of renal cell carcinoma with clear-cell component histology.
3. Locally advanced/metastatic renal cell carcinoma
4. Measurable lesion (RECIST 1.1) on physical exam or as CT/MRI
5. No prior systemic therapy for advanced/metastatic RCC
6. Karnofsky performance scale >=70
7. Age >=18 years
8. A female is eligible to enter and participate in this study if she is of: non-childbearing/agrees to use adequate contraception
9. A male with female partner of childbearing potential must have vasectomy/agree to use effective contraception from two weeks prior to administration of the 1st dose of study treatment for a period of time after the last dose of study treatment
10. Adequate organ function
11. Able to swallow and retain orally administered medication and must not have clinically significant GIT abnormalities that may alter absorption
12. The date of disease progression must be within six months of stopping sunitinib or during treatment with sunitinib
13. Measurable lesion at pazopanib baseline as per the RECIST 1.1 criteria

Exclusion Criteria:

1. Pregnant/lactating
2. History of another malignancy (unless have been disease-free for 3 years)
3. History or clinical evidence of Central nervous system metastases (unless have previously-treated CNS metastases and who meet both of the following criteria: a) are asymptomatic and b) have no requirement for steroids or enzyme-inducing anticonvulsants in prior 6 month time interval.
4. Clinically significant gastrointestinal abnormalities including, but not limited to: malabsorption syndrome, major resection of the stomach or small bowel that could affect the absorption of study drug, active peptic ulcer disease, known intraluminal metastatic lesion/s with suspected bleeding, Inflammatory bowel disease, ulcerative colitis, or other gastrointestinal conditions with increased risk of perforation, history of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess
5. Moderate to severe hepatic impairment (Child-Pugh Class C)
6. Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with patient's safety, obtaining informed consent or compliance to the study.
7. Subjects receiving chronic treatment with corticosteroids/other immunosuppressive agents
8. Subjects with a known history of HIV seropositivity
9. Subjects with active bleeding, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin)
10. Presence of any severe or uncontrolled medical conditions/infection.
11. Currently receiving chemotherapy, immunotherapy or radiotherapy
12. Corrected QT interval (QTc) > 480 milliseconds
13. History of any one or more of the following cardiovascular conditions within the past 12 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association
14. Poorly controlled hypertension (defined as systolic blood pressure of >=140mmHg or diastolic blood pressure of >=90mmHg).
15. History of cerebrovascular accident including transient ischemic attack, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months (unless recent DVT have been treated with therapeutic anti-coagulating agents for at least 6 weeks)
16. Major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer.
17. Evidence of active bleeding or bleeding susceptibility.
18. Known endobronchial lesion and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | pazopanib treatment until earliest date of disease progression or death, assessed up to 30 months after the last patient has been enrolled

SECONDARY OUTCOMES:
Overall survival of patients treated with second-line pazopanib therapy | Initiation of pazopanib dose until death, assessed up to 30 months after the last patient has been enrolled
Objective Response Rate to pazopanib therapy | Initiation of pazopanib treatment until time of confirmed best response, assessed up to 30 months after the last patient has been enrolled
Number of grade 3 or 4 adverse events attributable to pazopanib | Time of first dose of pazopanib to approximately one month after discontinuation of pazopanib

CONTACTS AND LOCATIONS:
Overall Officials: Mian Xie, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China